CLINICAL TRIAL: NCT05201365
Title: A Prospective Cohort Study of Compound Nanxing Zhitong Ointment in the Treatment of Chronic Musculoskeletal Pain
Brief Title: A Prospective Cohort Study of Compound Nanxing Zhitong Ointment
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Jiangsu Kanion Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: Z-FFNX-20211019-01
Record Dates: First submitted 2021-12-13; First posted 2022-01-21 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Chronic Musculoskeletal Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to evaluate the safety and the efficacy of compound Nanxing pain relief cream in the treatment of chronic pain in the musculoskeletal system

DETAILED DESCRIPTION:
Chronic pain, especially in the musculoskeletal system, is prevalent worldwide. Many studies show the burdens they impose: pain, disability, reduced quality of life (QoL), marked impairment of participation in work and social activities, and heavy financial costs.The purpose of this study is to evaluate the safety and the efficacy of compound Nanxing pain relief cream in the treatment of chronic pain in the musculoskeletal system. To provide a safe and effective treatment of Chronic Musculoskeletal Pain.

ELIGIBILITY:
Inclusion Criteria:

* Attendance at orthopedic, rheumatology and pain clinics for.

Exclusion Criteria:

* Indication for surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1. pain that meets the ICD-11 classification of chronic pain that is localized to the musculoskeletal system and occurs in the neck, shoulder, low back and extremities.
  2. Those who meet the criteria of "cold" in Chinese medicine and whose chronic pain is exacerbated by cold.
  3. Persistent/intermittent pain for more than 3 months and no indication for surgery.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Change in Overall Pain Assessment Scale score at week 12 overall Pain Assessment Scale score at week 12. | Change from Baseline GPS at week 12.
  Evaluation using Global pain scale, GPS。The change of pain assessment scale score from the beginning period of the treatment to the end indicates the effectiveness of the treatment.
  The GPS is based on patients' subjective and objective perceptions, and is used to measure patients' overall perceptions of pain. The scores were distributed from 0 to 10, with 0 representing no pain at all and 10 representing the most painful, and the scores were summarized and tallied. Higher scores indicate more severe pain effects.

SECONDARY OUTCOMES:
Quality of Life Short Form12,SF-12 | Total scores at baseline, week 2, week 4, week 8, and week 12 were evaluated in both groups.
  SF-12 The raw scores of the 7 dimensions were calculated separately. The scores ranged from 0 to 100, with 0 being the worst and 100 being the best.
Pain resolution time | VAS is assessed within 1 hour ahead of the treatment and within 1 hour after the treatment. The change of the score indicate the treatment efficacy.
  Visual analog scale(VAS) is used to test the painful degree. The time taken for a pain VAS score of ≤2 to be maintained for 24 hours or more.
Number of pain-free days per month | Records are taken every day by the end of the day. Records are assessed at the end of 12 weeks of treatment.
  Record the number of days per month that the patient is pain-free in the affected area.
Chinese medicine evidence score | The TCM evidence score was assessed within 1 hour after treatment. Changes in TCM evidence scores compared to baseline at week 12.
  The scale is divided into 2 main aspects, primary and secondary conditions. There are 2 entries for the primary condition. The secondary condition has 8 entries. The entries are scored as "0", "2", "4", and "6" depending on the severity of the symptoms. The total score is 36. The higher the score, the more severe the symptoms.
Safety evaluation | After 12 weeks of treatment, evaluate adverse reactions and make a record.
  Safety rating includes 4 levels.Level 1 means "Safe, without any adverse reactions".Level 2 means "Safer, if there is an adverse reaction, you can continue treatment without any treatment ".Level 3 means " Have safety problems, have moderate adverse reactions, and continue treatment after treatment". Level 4 means " Suspension test due to adverse reactions". Incidence of adverse events andadverse drug reactions.

CONTACTS AND LOCATIONS:
Overall Officials: chen weiheng, M.D., Study Chair — Vice President of the Third Affiliated Hospital of Beijing University of Chinese Medicine